CLINICAL TRIAL: NCT01237678
Title: A Phase 1/2 Study to Assess the Safety and Efficacy of Lorvotuzumab Mertansine in Combination With Carboplatin/Etoposide in Patients With Advanced Solid Tumors Including Extensive Stage Small Cell Lung Cancer
Brief Title: A Study of IMGN901 for Patients With Advanced Solid Tumors and Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped early due to lack of efficacy signal and safety concerns
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Immunogen 0007
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Small Cell Lung Cancer
Keywords: Immunogen; Lung; Small Cell Lung Cancer; Carboplatin; ADC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — lorvotuzumab mertansine; Carboplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMGN901 with carboplatin and etoposide (Experimental): Patients will receive IMGN901 along with carboplatin and etoposide for up to 6 cycles and then be able to continue on IMGN901 alone until no further benefit or toxicity.
  Interventions: Drug: IMGN901
- Carboplatin and Etoposide (Active Comparator): Patients will receive Carboplatin and etoposide for up to 6 cycles.
  Interventions: Drug: Carboplatin and Etoposide

INTERVENTIONS:
Drug: IMGN901 — Phase 2 regimen is IMGN901, Carboplatin, and Etoposide. IMGN901 to be given on days 1 and 8 every 21 days.
  Other Names: BB-10901, Lorvotuzumab mertansine
  Arms: IMGN901 with carboplatin and etoposide
Drug: Carboplatin and Etoposide — Patients assigned to Arm 2 were to receive carboplatin at the same AUC as utilized in Arm 1
  Other Names: Toposar®, VePesid®, Etopophos®
  Arms: Carboplatin and Etoposide

SUMMARY:
The purpose of this study is to test safety and efficacy of this combination treatment (IMGN901, carboplatin and etoposide) in patients with solid tumors and extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
Small-Cell Lung Cancer (SCLC) is a neuroendocrine cancer of the lung that is typically caused by smoking. Patients generally present with symptoms of cough, dyspnea, pain and weakness, and often have extensive disease at that time. It is estimated that 13% of lung cancers are SCLC in origin1. Approximately 28,530 new cases of SCLC were expected in 2009 based on an estimate of 219,440 new cases of any cancer of the lung in the US in 20092.

There are 2 stages of the disease: limited-stage disease (LD) and extensive-stage disease (ED). SCLC-LD is confined to a region of the chest (the hemithorax and mediastinum) that is more amenable to radiation therapy. Thirty percent (30%) of patients present with SCLC-LD. The remaining patients (70%) present with SCLC-ED, in which the disease has progressed outside this region of the chest. Common sites of metastatic disease include the contralateral lung, liver, adrenal glands, brain, bones and/or bone marrow3. Recurrence after therapy is typical. In the rare patient who has longer-term survival, secondary malignancies (new SCLC tumors and other malignancies) are common because of long-term exposure to carcinogens.

SCLC is very responsive to chemotherapy and radiation therapy, having response rates of up to 80%4-7. In limited stage disease, the standard treatment is 'combined-modality therapy' consisting of combination chemotherapy such as cisplatin plus etoposide followed by thoracic radiation therapy. Surgery is rarely used.

Despite high response rates, therapy is rarely curative due to high rates of recurrence and metastasis. Overall 5-year survival for SCLC patients is 4%5. SCLC-LD patients typically achieve median survival of 14 to 24 months after therapy, with a 2-year survival rate of 40% to 50%. This survival rate drops to about 20% at 5 years4-7. SCLC-ED patients achieve a median survival of 8 to 12 months on therapy8.

Patients will typically have recurrent disease after therapy. While many of these patients may be eligible for further chemotherapy, survival at this stage is usually less than 6 months.

No treatment modality has a significant impact on overall survival. Studies utilizing regimens with greater numbers of chemotherapeutic agents or longer therapy duration have not improved survival. Thus, a new therapy that can improve survival is needed.

IMGN901 is an antibody drug conjugate which is anticipated to result in lower systemic toxicity and greater efficacy than currently available therapies based on its specific and high affinity binding to its target antigen, CD56. This antigen has been shown to be present in almost all cases of SCLC (~ 95% based on in-house data). In in vivo studies, IMGN901 has demonstrated potent anti-tumor activity against CD56-positive carcinomas including xenograft models of SCLC as well as complete regressions when combined with cisplatin/etoposide. Preliminary clinical activity of single agent IMGN901 based on data from two Phase 1 studies shows a disease control rate (PR and SD, defined as non-progression for at least 75 days) estimated to be 24% in a heterogeneous population of patients with pretreated and drug resistant SCLC. Additional data supportive of the potential activity of IMGN901 includes complete responses and clinically relevant stable disease in patients with MCC (clinical benefit rate = 39%). Further, the tolerability profile demonstrating minimal myelosuppression with administration of IMGN901 is supportive of exploring its use in combination with established chemotherapy regimens.

IMGN901 is supportive of exploring its use in combination with established chemotherapy regimens.

Therefore, the Phase 1 portion of this study is designed to first determine the MTD, presumably the recommended Phase 2 dose, of IMGN901 when administered in combination with carboplatin/etoposide treatment and to characterize the safety, tolerability, PK, pharmacodynamics, immunogenicity, and preliminary anti-tumor activity of this triplet combination.

Improvement in disease control and survival of patients with SCLC-ED remains a major therapeutic challenge. New agents with better activity and tolerability are needed for this population. However, because large-scale clinical studies often are necessary to demonstrate the safety and effectiveness of these new agents, it is desirable to first evaluate some measure of relative effectiveness in a Phase 2 study.

Therefore the Phase 2 portion of the study will utilize a Simon two-stage design in which the activity of IMGN901 will be assessed by comparing the PFS rate at six months in the IMGN901 experimental arm (triplet combination) against the historical 6 month PFS rate of 0.44 (equivalently a median PFS = 5 months). In this study, an improvement of 2.5 months in median PFS will be deemed clinically relevant and correlates to a PFS rate of 0.58 (HR = 0.667). The control arm will be used primarily to reliably assess the safety of IMGN901 and will further serve as an informal validation of the historical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years old
* Patients must have been diagnosed with small-cell lung cancer (SCLC) and extensive disease
* ECOG performance status of 0, 1, or 2
* No prior systemic chemotherapy for the treatment of SCLC

Exclusion Criteria:

- Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (32):
  - Arizona Cancer Center @ UMC North, Tucson, Arizona
  - UCLA Oncology Center, Los Angeles, California
  - St. Joseph's Hospital, Orange, California
  - UCLA Hematology, Pasadena, California
  - UCLA Oncology Clinic, Santa Monica, California
  - UCLA Santa Clarita Valley Cancer Center, Valencia, California
  - UCLA Oncology Center, Westlake Village, California
  - Yale Medical Center, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Johnson Therurer Cancer Center at Hackensack, Hackensack, New Jersey
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Cancer Centers East, Oxford Drive, Monroeville, Pennsylvania
  - UPMC Cancer Center St. Margaret, Pittsburgh, Pennsylvania
  - Univeristy of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant (HOA), Pittsburgh, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UTHSC at San Antonio, San Antonio, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Canada (5):
  - Juravinski Cancer Center, Hamilton, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
  - Royal Victoria, Montreal, Quebec
- Spain (6):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu y Sand Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (5):
  - Royal Sussex Hospital, Brighton, East Sussex
  - University College of London, London, England
  - The Christie Hospital, Withington, Manchester
  - Royal Marsden, Sutton, Surrey
  - Royal Marsden, London, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from, and treated at, 45 study sites in the U.S., Canada, Spain, and the U.K. between November 2010 and May 2015.
Pre-assignment Details: Patients were screened during a 28-day period
Groups:
- Phase I - IMGN901 + Carboplatin + Etoposide: Participants received IMGN901 on Days 1 and 8 of a 21-day cycle. All patients also received carboplatin on Day 1 and etoposide on Days 1, 2, and 3 of each 21-day cycle.The starting dose of IMGN901 was 60 mg/m2; dose escalation proceeded, as tolerated, through 75, 90, and 112 mg/m2. Carboplatin was originally dosed at an AUC 6 however due to poor tolerability this was reduced to an AUC of 5. Study drug combinations were administered for four cycles, with up to 6 cycles allowed. IMGN901 was continued as monotherapy for patients who achieved a response or stable disease.
- Phase II - IMGN901 + Carboplatin + Etoposide: IMGN901 was administered at the RP2D (recommended phase II dose) determined in Phase I (112 mg/m2; later reduced to 90 mg/m2) on Days 1 and 8 of each 21-day cycle. Patients also received carboplatin (AUC 5) on Day 1 and etoposide (100 mg/m2) on Days 1, 2, and 3 of each 21-day cycle. Study drug combinations were administered for four cycles, with up to 6 cycles allowed. IMGN901 was continued as monotherapy for patients who achieved a response or stable disease.
- Phase II - Carboplatin + Etoposide: Carboplatin (AUC 5) was administered on Day 1 and etoposide (100 mg/m2) on Days 1, 2, and 3 of each 21-day cycle. Drugs were administered for 6 cycles as tolerated.
Period: Phase I - IMGN901+Carboplatin+Etoposide
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide
Started | 33 | 0 | 0
Received Intervention | 33 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 33 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lack of Efficacy | 24 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Incorrect Original Diagnosis | 1 | 0 | 0
Period: Phase II
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide
Started | 0 | 98 (98 subjects were randomized, 94 subjects treated) | 50 (50 subjects were randomized, 47 subjects treated)
Received Intervention | 0 | 94 | 47
Completed | 0 | 0 | 0
Not Completed | 0 | 98 | 50
Not completed — Adverse Event | 0 | 39 | 9
Not completed — Death | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 25 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 5
Not completed — Completed Cycles 4-6 | 0 | 11 | 21
Not completed — Sponsor Decision/Study Closed | 0 | 18 | 7
Not completed — Randomized but were not treated | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Phase II - IMGN901 + Carboplatin + Etoposide: IMGN901 was administered at the RP2D determined in Phase I (112 mg/m2; later reduced to 90 mg/m2) on Days 1 and 8 of each 21-day cycle. Patients also received carboplatin (AUC 5) on Day 1 and etoposide (100 mg/m2) on Days 1, 2, and 3 of each 21-day cycle. Study drug combinations were administered for four cycles, with up to 6 cycles allowed. IMGN901 was continued as monotherapy for patients who achieved a response or stable disease.
- Total: Total of all reporting groups
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide | Total
Number analyzed (Participants) | 33 | 94 | 47 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 49 | 26 | 96
  >=65 years | 12 | 45 | 21 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 40 | 22 | 82
  Male | 13 | 54 | 25 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 7
  White | 30 | 90 | 44 | 164
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0 = Fully active, able to carry out all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. = Ambulatory and capable of all self-care but unable to carry out work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 14 | 22 | 12 | 48
    1 | 19 | 62 | 32 | 113
    2 | 0 | 10 | 3 | 13
History of Smoking [Number; unit: participants]
  Yes | 21 | 93 | 46 | 160
  No | 12 | 1 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Dose Limiting Toxicities (DLT)
Description: The primary outcome measure for Phase I was to determine the maximum tolerated dose (MTD) and characterize the dose limiting toxicities (DLT) of IMGN901 when administered in combination with carboplatin/etoposide chemotherapy followed by IMGN901 alone in patients with solid tumors. For the purposes of dose escalation and determination of MTD, DLTs were defined as AEs or abnormal laboratory values related to study treatment which occurred in Cycle 1 of the Dose Escalation phase, including any AEs that resulted in failure to meet the criteria for re-treatment. The following events were considered DLTs (using the most current version of CTCAE): febrile neutropenia; Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding; ≥ Grade 3 peripheral neuropathy; ≥ Grade 3 vomiting, nausea, or diarrhea that persisted despite the use of optimal therapy; other ≥ grade 3 non-hematologic toxicity (with the exception of brief fatigue i.e. ≤ 72 hours and alopecia)
Time Frame: 21 days (Cycle 1)
Population: A total of 33 patients were analyzed as part of the Dose escalation phase.
Measure: Number; unit: participants
Arm/Group | IMGN901 60 mg/m2 + Carboplatin AUC 6 + Etoposide 100 mg/m2 | IMGN901 75 mg/m2 + Carboplatin AUC 6 + Etoposide 100 mg/m2 | IMGN901 75 mg/m2 + Carboplatin AUC 5 + Etoposide 100 mg/m2 | IMGN901 90 mg/m2 + Carboplatin AUC 5 + Etoposide 100 mg/m2 | IMGN901 112 mg/m2 + Carboplatin AUC 5 + Etoposide 100 mg/m2
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 12
participants
  Grade 3 febrile neutropenia | 0 | 1 | 0 | 0 | 0
  Grade 4 febrile neutropenia | 1 | 1 | 0 | 1 | 0
  Grade 4 thrombocytopenia | 0 | 2 | 0 | 1 | 1
  Grade 4 granulocytopenia | 0 | 1 | 0 | 0 | 0
  Grade 3 lobar pneumonia | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Progression Free Survival (PFS) in Phase II
Description: The primary outcome measure for Phase II was to determine the efficacy of IMGN901 in combination with carboplatin/etoposide chemotherapy as first-line treatment for patients with extensive stage small cell lung cancer. PFS was defined as the time from enrollment until objective tumor progression according to RECIST 1.1 or death on study due to any cause, whichever occurred first. Only the results from the experimental arm (IMGN901 + carboplatin + etoposide) are presented as the primary objective of this phase of the study was to compare PFS in the experimental arm (triplet combination) against historical PFS rates for carboplatin and etoposide. The control arm was planned primarily to reliably assess the safety of IMGN901 and to demonstrate whether the or not the historical assumptions regarding efficacy were confirmed.
Time Frame: From randomization to objective tumor progression or death (up to post-treatment follow-up 28 days after last dose, up to 22 months)
Population: A total of 82 patients from the IMGN901 + carboplatin + etoposide safety population (N=94) were included in the efficacy analyses, due to the lack of post-baseline evaluations for 12 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II - IMGN901 + Carboplatin + Etoposide
Number analyzed (Participants) | 82
months | 6.2 [5.4 to 7.2]

3. Primary Outcome: Maximum Tolerated Dose (MTD) of IMGN901
Description: A primary outcome measure for Phase I was to determine the maximum tolerated dose (MTD) of IMGN901 when administered in combination with carboplatin/etoposide chemotherapy followed by IMGN901 alone in patients with solid tumors. The MTD was determined based on DLTs that occurred during Cycle 1.
Time Frame: 21 days (Cycle 1)
Population: During escalation, carboplatin dosing was reduced from AUC 6 to AUC 5 due to poor tolerability; therefore the MTD for IMGN901 was determined in combination with carboplatin AUC5 and 100 mg/m^2 etoposide
Measure: Number; unit: mg/m^2
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide
Number analyzed (Participants) | 33
mg/m^2 | 112

4. Secondary Outcome: Overview of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: To assess the type and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs). An AE was defined as any noxious, pathologic, or unintended change un anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of the study, whether or not deemed study drug-related. An SAE was any AE resulting in death, life-threatening experience, initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, or congenital defect. All AEs were reported from the time of the first dose of study treatment until 28 days after the final dose of study drug. the severity of AEs were graded by the Investigator using National cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) version 4.0.
Time Frame: From the first dose of study drug on Cycle 1, Day 1 until 28 days after the last study treatment (up to 22 months)
Measure: Number; unit: participants
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide
Number analyzed (Participants) | 33 | 94 | 47
participants
  Any TEAE | 33 | 94 | 46
  Related TEAE | 32 | 90 | 39
  Any SAE | 16 | 54 | 23
  Related SAE | 8 | 30 | 9
  TEAEs leading to discontinuation | 8 | 50 | 6
  Any Grade ≥ 3 TEAE | 29 | 92 | 42
  Related Grade ≥ 3 TEAE | 22 | 83 | 33
  Deaths within 28 days of last dose | 1 | 14 | 5

5. Secondary Outcome: Progression Free Survival (PFS) Rate at 6 Months
Description: The trial was not empowered to permit a statistically informative comparison of the randomized treatment groups with respect to PFS. The activity of IMGN901 was assessed by comparing the PFS rate at 6 months in the IMGN901 experimental arm against the historical 6-month PFS rate of 0.44 (equivalently a median PFS = 5 months). Only the results from the experimental arm (IMGN901 + carboplatin + etoposide) are presented as the objective was to compare PFS at 6 months in the experimental arm (triplet combination) against the historical PFS rate of 0.44 (equivalently a median PFS = 5 months) for carboplatin and etoposide. The control arm was planned primarily to reliably assess the safety of IMGN901 and to demonstrate whether the or not the historical assumptions regarding efficacy were confirmed.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II - IMGN901 + Carboplatin + Etoposide
Number analyzed (Participants) | 82
percentage of participants | 39 [28.4 to 50.4]

6. Secondary Outcome: Median Overall Survival (OS) in Phase II
Description: A secondary outcome measure for Phase II was to determine the overall survival of patients treated with IMGN901 in combination with carboplatin/etoposide chemotherapy versus carboplatin/etoposide chemotherapy alone as first-line treatment for patients with extensive stage small cell lung cancer.
Time Frame: From the time of enrollment until death on study due to any cause (up to post-treatment follow-up 28 days after last dose, up to 22 months)
Population: A total of 121 patents were included in the analyses (82 in Arm1 and 39 in Arm 2) due to due to the lack of post-baseline evaluations for 20 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide
Number analyzed (Participants) | 82 | 39
months | 10.1 [8.7 to 18.1] | 10.97 [7.5 to 11.4]

7. Secondary Outcome: Overall Survival (OS) Rate at 12 Months
Description: OS was analyzed based on a binary definition of the number of patients dead or censored prior to 12 months and the number of patients alive at 12 months. The primary objective of this phase of the study was to compare PFS in the experimental arm (triplet combination) against historical PFS rates. The control arm was primarily planned to demonstrate whether the or not the historical assumptions regarding efficacy were confirmed. Further, the trial was not empowered to permit a statistically informative comparison of the randomized treatment groups with respect to OS and no determination of the OS rate at 12 months for the control arm was performed; therefore only the results from the experimental arm (IMGN901 + carboplatin + etoposide) are presented.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants alive
Arm/Group | Phase II - IMGN901 + Carboplatin + Etoposide
Number analyzed (Participants) | 82
percentage of participants alive | 61 [49.6 to 71.6]

ADVERSE EVENTS:
Time Frame: Reported SAEs include events from the first dose of study drug on Cycle 1, Day 1 until 28 days after the last study treatment.
Description: AEs and laboratory results were graded using the NCI CTCAE, version 4.0.
Groups:
- Phase I - IMGN901 + Carboplatin + Etoposide: Participants received IMGN901 on Days 1 and 8 of a 21-day cycle. All patients also received carboplatin on Day 1 and etoposide (100 mg/m2) on Days 1, 2, and 3 of each 21-day cycle. The starting dose of IMGN901 was 60 mg/m2; dose escalation proceeded, as tolerated, through 75, 90, and 112 mg/m2. Carboplatin was originally dosed at an AUC 6 however due to poor tolerability this was reduced to an AUC of 5. Study drug combinations were administered for four cycles, with up to 6 cycles allowed. IMGN901 was continued as monotherapy for patients who achieved a response or stable disease.
Arm/Group | Phase I - IMGN901 + Carboplatin + Etoposide | Phase II - IMGN901 + Carboplatin + Etoposide | Phase II - Carboplatin + Etoposide
Serious Adverse Events (participants affected / at risk) | 16/33 | 54/94 | 23/47
Other Adverse Events (participants affected / at risk) | 33/33 | 91/94 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - IMGN901 + Carboplatin + Etoposide (N=33) | Phase II - IMGN901 + Carboplatin + Etoposide (N=94) | Phase II - Carboplatin + Etoposide (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Atrial defibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2 | 0
Pain (General disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Disease progression (General disorders) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 4 | 1
Pneumonia (Infections and infestations) | 0 | 6 | 2
Sepsis (Infections and infestations) | 2 | 2 | 1
Septic shock (Infections and infestations) | 0 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0
Vulval haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal heamorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal heamorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - IMGN901 + Carboplatin + Etoposide (N=33) | Phase II - IMGN901 + Carboplatin + Etoposide (N=94) | Phase II - Carboplatin + Etoposide (N=47)
Anaemia (Blood and lymphatic system disorders) | 24 | 50 | 21
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 10 | 6
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 53 | 24
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 32 | 19
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 3
Constipation (Gastrointestinal disorders) | 12 | 30 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 30 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 13 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 4
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 40 | 17
Vomiting (Gastrointestinal disorders) | 11 | 23 | 11
Asthenia (General disorders) | 3 | 29 | 10
Chills (General disorders) | 2 | 6 | 2
Fatigue (General disorders) | 17 | 46 | 14
Influenza like illness (General disorders) | 2 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 13 | 6
Oedema peripheral (General disorders) | 3 | 19 | 5
Pain (General disorders) | 5 | 7 | 2
Pyrexia (General disorders) | 8 | 10 | 5
Oral candidiasis (Infections and infestations) | 3 | 5 | 2
Urinary tract infection (Infections and infestations) | 5 | 10 | 7
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 11 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 8 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 8 | 1
Blood creatine increased (Investigations) | 3 | 2 | 3
Blood pressure increased (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0
Lipase increased (Investigations) | 2 | 3 | 3
Lymphocyte count decreased (Investigations) | 7 | 0 | 0
Neutrophil count decreased (Investigations) | 7 | 11 | 7
Platelet count decreased (Investigations) | 2 | 16 | 6
Weight decreased (Investigations) | 2 | 7 | 3
White blood cell count decreased (Investigations) | 7 | 8 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 32 | 16
Dehydration (Metabolism and nutrition disorders) | 3 | 15 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 13 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 16 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 12 | 6
Hypophospataemia (Metabolism and nutrition disorders) | 5 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 18 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 12 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 11 | 3
Dizziness (Nervous system disorders) | 3 | 13 | 5
Dysgeusia (Nervous system disorders) | 4 | 10 | 6
Headache (Nervous system disorders) | 7 | 16 | 5
Paraesthesia (Nervous system disorders) | 2 | 20 | 2
Peripheral motor neuropathy (Nervous system disorders) | 2 | 7 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 56 | 4
Restless legs syndrome (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 8 | 1
Depression (Psychiatric disorders) | 2 | 5 | 1
Insomnia (Psychiatric disorders) | 6 | 19 | 4
Dysuria (Renal and urinary disorders) | 4 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 18 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 32 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 2 | 7 | 0
Hypotension (Vascular disorders) | 2 | 10 | 4
Sinus tachycardia (Cardiac disorders) | 0 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 6 | 2
Malaise (General disorders) | 0 | 6 | 0
Non-cardiac chest pain (General disorders) | 0 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 2
Blood amylase increased (Investigations) | 0 | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 12 | 3
Hyporeflexia (Nervous system disorders) | 0 | 0 | 3
Neurotoxicity (Nervous system disorders) | 0 | 8 | 1
Hot flush (Vascular disorders) | 0 | 5 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days